CLINICAL TRIAL: NCT05443854
Title: Impact of Aminoglycosides-based Antibiotics Combination and Protective Isolation on Outcomes in Critically-ill Neutropenic Patients With Sepsis: A Randomized 2 by 2 Factorial Design Randomized Pragmatic Trial.
Brief Title: Impact of Aminoglycosides-based Antibiotics Combination and Protective Isolation on Outcomes in Critically-ill Neutropenic Patients With Sepsis: (Combination-Lock01)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: APHP180690
Record Dates: First submitted 2022-06-17; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Sepsis; Septic Shock; Hematologic Malignancy; Tumor; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Sepsis; Shock, Septic; Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aminoglycosides intervention (Experimental): Systematic aminoglycoside therapy using Amikacin at a dose of 25 to 30 mg/Kg per dose, at a rate of a maximum of 1 infusion per day will be delivered.
  Recommended duration will be of three days or until microbiological documentation.
  Interventions: Drug: Aminoglycosides intervention
- Lack of protective isolation intervention (Experimental): Protective isolation will be avoided until ICU discharge is deemed possible. Specific measures regarding nutrition (including avoidance of food consider at risk of fungal contamination) and water protection will be maintained.
  Interventions: Behavioral: Lack of protective isolation intervention
- No systematic aminoglycosides intervention (Other): Antibiotic therapy and prophylaxis will be in line with more recent IDSA and ESCMID guidelines - standard arm
  Interventions: Other: No systematic aminoglycosides intervention - standard arm
- Protective isolation intervention (Other): Protective isolation will be provided systematically as currently practiced in participating centers - standard arm
  Interventions: Other: Protective isolation intervention - standard arm

INTERVENTIONS:
Drug: Aminoglycosides intervention — Antibiotic therapy and prophylaxis will be in line with more recent IDSA and ESCMID guidelines [3, 28, 50].
  Systematic aminoglycoside therapy using Amikacin at a dose of 25 to 30 mg/Kg per dose, at a rate of a maximum of 1 infusion per day will be delivered.
  Recommended duration will be of three days or until microbiological documentation.
  Arms: Aminoglycosides intervention
Behavioral: Lack of protective isolation intervention — Protective isolation will be avoided until ICU discharge is deemed possible. Specific measures regarding nutrition (including avoidance of food consider at risk of fungal contamination) and water protection will be maintained.
  Extended universal hygiene measures will be maintained and use of mask will be advocated during viral epidemic periods.
  A high degree of compliance as regard to antifungal prophylaxis guidelines and local standard hygiene procedures will be advocated
  Arms: Lack of protective isolation intervention
Other: No systematic aminoglycosides intervention - standard arm — Antibiotic therapy and prophylaxis will be in line with more recent IDSA and ESCMID guidelines [3, 28, 50].
  No systematic aminoglycoside therapy will be provided except in presence of predefined specific organ infection (such intra-vascular infection such endocarditis for example) or drug-resistant infection requiring aminoglycosides.
  Arms: No systematic aminoglycosides intervention
Other: Protective isolation intervention - standard arm — Protective isolation will be provided systematically as currently practiced in participating centers. Modality will be in line with recent SRLF guidelines, we will recommend for the patients to receive an isolation the maximal available isolation with the aim to provide:
  1. High-efficiency air filtration [filtration of 99.7% of particles greater than or equal to 0.3 µm; International Organization for Standardization (ISO) class 5 or better]
  2. Geographical isolation in an individual room
  3. Technical isolation, including a face mask and a cap. This approach of isolation will however be pragmatic on the basis of the "best available" level of isolation in line with recommendation, while not delaying ICU admission and patients' care
  Arms: Protective isolation intervention

SUMMARY:
Sepsis remains the leading cause of ICU admission in neutropenic patients. This condition remains associated with a high morbidity and mortality, with hospital mortality of 60% when vasopressors are required.

Full protective isolation (including geographic isolation, technical isolation, high-efficiency air filtration, and digestive decontamination) proved to be efficient in patients with profound and prolonged neutropenia with regard to infection rate. However, these studies are biased and were performed up to 40 years ago. More recent studies, performed in patients with less profound neutropenia, or performed without digestive decontamination or with partial protective isolation led however to negative results. More importantly, isolation has been demonstrated to limit access to patients' room and to be associated with suboptimal monitoring, with increased rate of severe and avoidable adverse events. This may explain the uneven use of protective isolation in hematology ward and expert's suggestion to appraise protective isolation benefits using large well conducted RCT.

In neutropenic patients with suspected sepsis, urgent broad antibiotic therapy is mandatory and failure to initiate adequate antibiotic therapy within 1 hour has been associated with a 10 fold increase in adjusted mortality. Current IDSA guidelines recommend using preferentially large anti-pseudomonas beta-lactam therapy. Routine antibiotic combination using aminoglycosides is controversial and not recommended. On one hand, meta-analyses suggested not-only a lack of benefit from this association but also increased rate of renal failure and a trend towards a higher mortality rate with aminoglycosides use. On the other hand, subgroup analysis and low-level evidences studies suggest however a benefit from aminoglycosides in critically-ill patients, patients with severe sepsis, or those with documented gram negative infection. Along this line, both the recent Cochran systematic review and the recent French guidelines focusing on neutropenia management in critically-ill patients advocated additional trials in this field focusing in the sickest patients.

The current study aims to assess benefits of protective isolation and systematic use of aminoglycosides combination antibiotic therapy in critically-ill patients with cancer-related neutropenia and sepsis or septic shock. To do so, the investigators intend to perform a 2x2 factorial design randomized pragmatic trial comparing on one hand benefits of protective isolation (versus no protective isolation) and in the other hand benefits of systematic aminoglycosides antibiotics combination (versus no systematic combination).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Sepsis or septic shock as defined by SEPSIS3 definition
* Underlying tumor, allogeneic stem cell transplantation or hematological malignancy
* Neutropenia (defined by either absolute neutrophil count <500/mm3 or leucocytes <1000/mm3) related to an underlying malignancy or its treatment
* Informed or deferred consent

Exclusion Criteria:

* Pregnancy and breastfeeding
* Moribund patients (death expected within 48 hours by attending physician)
* Previous participation to this study
* No affiliation to social security
* Patients under legal protection according to French Law
* Patient having received more than 1 injection of aminoglycosides in the 3 days preceding ICU admission
* Contraindication to aminoglycosides as mentioned in SpC section 4.3:

  * Hypersensitivity to amikacin, to other antibiotics from the aminoglycoside family, or to any excipient from the amikacin used.
  * Patients with documented allergy to aminoglycosides
  * Myasthenia gravis
  * Concomitant administration of intravenous Polymyxin- Delay between admission for a new sepsis and inclusion>24 hours or (in patients previously admitted in the ICU for another reason) delay between new sepsis in study inclusion >24h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Mortality | at day 90
  Overall death

SECONDARY OUTCOMES:
Mortality | at Day-28
  Overall death
Hospital mortality | at hospital discharge within 3 months
  Mortality at hospital discharge
Incidence of acute kidney injury | within 3 months
  Acute kidney injury (AKI) will be defined according to KDIGO criteria
Severity of acute kidney injury | within 3 months
  Acute kidney injury (AKI) will be defined according to KDIGO criteria
Duration of acute kidney injury | within 3 months
  Acute kidney injury (AKI) will be defined according to KDIGO criteria
Major Adverse Kidney Events | at day-28
Major Adverse Kidney Events | at day 90
Incidence of clinically apparent loss of hearing | at ICU discharge
Incidence of clinically apparent loss of hearing | at dat 90
Rate of adherence of hand hygiene | at 24 hours
  hand hygiene will be assessed by external observer
Incidence density of selected serious adverse events | within 3 months
Incidence density of new bacterial episodes | within 3 months
Incidence density of new viral infection episodes | within 3 months
Incidence density of new fungal episodes | within 3 months
Number of days free from organ support therapy (mechanical ventilation, vasopressors or RRT) | at day 28
Rate of clinical cure | within 3 months
Frequency of initial antibiotic therapy inadequate as regard to microbiological documentation. | at inclusion
Number of day free of antibiotic therapy | at day-28
Duration of aminoglycoside therapy | within 3 months
Rate of aminoglycoside overdosage according to residual concentration | within 3 months
Rate of overuse when compared to experts recommendations | within 3 months

IPD SHARING:
Plan to Share IPD: Undecided